CLINICAL TRIAL: NCT03217721
Title: Antibiotics Management of Septic Neutropenic Patients in the Intensive Care Unit : New Recommendations do They Change Our Clinical Practice ?
Brief Title: Antibiotics Management of Septic Neutropenic Patients in the Intensive Care Unit
Acronym: REANEUF
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC17.0092 - REANEUF
Record Dates: First submitted 2017-07-05; First posted 2017-07-14 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2017-07

CONDITIONS: Neutropenia, Febrile
MeSH Terms: conditions — Febrile Neutropenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neutropenia, defined by an absolute count of polymorphonuclear neutrophils less than <1500/mm3, exposes patients to infectious complications that can lead to sepsis or septic shock. The mortality risk is higher risk. The recommendations published in 2016 were formulated to homogenize the clinical practices to improve the survival.

DETAILED DESCRIPTION:
We evaluate the adequacy antibiotics prescriptions in febrile neutropenia with suspected infection and evaluate factors influencing adequacy therapy and mortality consequence.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis or septic shock at admission or during the stay

Exclusion Criteria:

* Minor
* Pregnancy
* Opposition

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Pilot, exploratory, monocentric, retrospective, observational study
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
Proportion of adequate antibiotic prescription | Through study completion, an average of 1 month
  Proportion of adequate antibiotic prescription

SECONDARY OUTCOMES:
Mortality of all causes | ICU, hospital and 28-day mortality
  Mortality of all causes

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schnell D, Azoulay E, Benoit D, Clouzeau B, Demaret P, Ducassou S, Frange P, Lafaurie M, Legrand M, Meert AP, Mokart D, Naudin J, Pene F, Rabbat A, Raffoux E, Ribaud P, Richard JC, Vincent F, Zahar JR, Darmon M. Management of neutropenic patients in the intensive care unit (NEWBORNS EXCLUDED) recommendations from an expert panel from the French Intensive Care Society (SRLF) with the French Group for Pediatric Intensive Care Emergencies (GFRUP), the French Society of Anesthesia and Intensive Care (SFAR), the French Society of Hematology (SFH), the French Society for Hospital Hygiene (SF2H), and the French Infectious Diseases Society (SPILF). Ann Intensive Care. 2016 Dec;6(1):90. doi: 10.1186/s13613-016-0189-6. Epub 2016 Sep 15. PMID 27638133